CLINICAL TRIAL: NCT00714441
Title: Reducing Distress and Improving Self-Care in Diabetes
Acronym: REDEEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2R01DK061937-05A1 (NIH); 2R01DK061937-05A1 (NIH)
Record Dates: First submitted 2008-07-09; First posted 2008-07-14 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Diabetes Type 2
Keywords: Diabetes Type 2; Distress; Problem Solving Therapy; Computer Automated Self-Management (CASM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2 (Active Comparator): Computer Automated Self-Management (CASM). Please see description below for CASM.
  Interventions: Behavioral: Computer Automated Self-Management (CASM)
- 3 (Active Comparator): Computer Automated Self-Management and Problem Solving Therapy (CAPS). Please see descriptions below for CAPS (also refer to CASM with is included in the CAPS program).
  Interventions: Behavioral: Computer Automated Self-Management (CASM); Behavioral: Computer Automated Self-Management and Problem Solving Therapy (CAPS)
- 1 (Active Comparator): Lifestyle and Activities Education Program (LEAP-AHEAD). Please see description below for LEAP-AHEAD.
  Interventions: Behavioral: Lifestyle and Activities Education Program (LEAP-AHEAD)

INTERVENTIONS:
Behavioral: Lifestyle and Activities Education Program (LEAP-AHEAD) — Patients in the LEAP-AHEAD Program arm will be shown a 40-minute interactional DVD and given the Healthy Habits Health Risk Appraisal, at baseline and 20 weeks that asks questions about diabetes self care practices and other health behaviors and gives recommendations in those areas. A score sheet based on the participant's responses will be left with the participant. At intervals from 0 to 44 weeks, patients will receive emailed informational pamphlets on diabetes and its complications, along with live telephone calls to answer any questions and check-in.
  Arms: 1
Behavioral: Computer Automated Self-Management (CASM) — CASM is a live and computer-assisted, low intensity, automated web and telephony based program that is directed at enhancing and sustaining diabetes self-management behavior over time. It provides education on the importance of healthy eating, physical activity and medication taking, and then asks patients to select an area for behavior change. At baseline patients will have a 45 minutes home visit to help them set goals and familiarize them with the website. A booster session is given at 20 weeks. Patients receive 8 ive phone calls over 12 months to support behavior change efforts.
  Arms: 2; 3
Behavioral: Computer Automated Self-Management and Problem Solving Therapy (CAPS) — Patients in the CAPS program receive all of the protocol included in the CASM program, and in addition receive a Problem Solving program. Problem solving is a process by which an individual attempts an adaptive solution to stressful, real life problem(s). At baseline there is a 45 minute home visit where the Counselor will introduce the patient to CASM and will go on to teach the patient about diabetes distress and PST. They will then generate a list of distress-related problems to teach the steps of PST. The steps of PST are: problem definition, goal setting, brain storming, decision making, action planning, and solution review. At 20 weeks there will be a booster session. Patients receive 8 live phone calls over 12 months to support behavior change efforts.
  Arms: 3

SUMMARY:
To date, there have been few practical, evidenced based interventions that are directed at patients with Type II Diabetes who are experiencing depressed and/or emotional distress in primary care settings. This study will (1) combine two existing, evidenced-based, interventions (a computer automated, diabetes specific self-management program (CASM) vs. a self-care program plus a live problem solving distress-reduction program (CAPS) vs. a lifestyle and activities education program (LEAP-AHEAD)) into a practical, 3-arm clinical trial with a highly distressed multi-ethnic patient sample, and (2) evaluate the intervention using the RE-AIM framework, sharing the results through a comprehensive dissemination package.

Hypothesis 1: The combined CASM and CAPS arms will be superior to the LEAP-AHEAD group on the primary outcomes at follow-up.

Hypothesis 2: The CAPS arm will be superior to the CASM arm on primary outcomes at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of type 2 diabetes (confirmed using the Wellborn criteria for a minimum of 12 months)
* Be between 21 and 75 years of age
* Speak and read Spanish or English fluently
* In addition, based on the telephone screening, patients will have to display a high level of diabetes distress and a deficit in at least one of three self-management areas (diet, physical activity, medication adherence). This is defined as having an average item score > 3.0 on 2 items from the regimen distress and emotional burden sub scale of the DDS and indication of problems in management on at least one scale of the SDSCA (i.e., endorsing having a healthy eating plan on less than 5 days/week, 30 minutes physical activity less than 5 days/week, or forget to take medicines more than 1 day/week).
* Have access to the internet

Exclusion Criteria:

* Have major disabilities or severe disorders (MI in the last 12 months, psychosis, on end-stage dialysis, dementia)
* Have current MDD (based on the PHQ8).

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2008-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Diet. Starting the Conversation is a 9 items measure of eating patterns (including 2 items from the NCI Fruit and Vegetable Screener). NCI Percent Energy from Fat Screen (PFAT) contains 17 items concerning frequency of intake for 15 food groups. | Baseline, 16 weeks, and 12 months
Physical Activity. The CHAMPS (28 items) will be used to measure physical activity. | Baseline, 16 weeks, and 12 months
Medication Adherence. Medication taking will be assessed by the Hill-Bone Medication Adherence scale. Questions will also cover smoking and alcohol use. | Baseline, 16 weeks, and 12 months
Distress. Patient distress will be assessed across several measures including: the 20-item CES-D, the 17-item DDS, the PHQ8, and screening items from the SCID to rule out psychosis. | Baseline, 16 weeks, and 12 months

SECONDARY OUTCOMES:
HbA1C | Baseline, 16 weeks, and 12 months
Blood Pressure | Baseline, 16 weeks, and 12 months
Fasting glucose | Baseline, 16 weeks, and 12 months
Lipids | Baseline, 16 weeks, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Fisher, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- UC San Francisco, Family and Community Medicine Dept., San Francisco, California, United States

REFERENCES:
- [Background] Fisher L, Glasgow RE, Mullan JT, Skaff MM, Polonsky WH. Development of a brief diabetes distress screening instrument. Ann Fam Med. 2008 May-Jun;6(3):246-52. doi: 10.1370/afm.842. PMID 18474888
- [Background] Fisher L, Skaff MM, Mullan JT, Arean P, Mohr D, Masharani U, Glasgow R, Laurencin G. Clinical depression versus distress among patients with type 2 diabetes: not just a question of semantics. Diabetes Care. 2007 Mar;30(3):542-8. doi: 10.2337/dc06-1614. PMID 17327318
- [Background] Glasgow RE, Fisher L, Skaff M, Mullan J, Toobert DJ. Problem solving and diabetes self-management: investigation in a large, multiracial sample. Diabetes Care. 2007 Jan;30(1):33-7. doi: 10.2337/dc06-1390. PMID 17192329
- [Background] Arean PA, Perri MG, Nezu AM, Schein RL, Christopher F, Joseph TX. Comparative effectiveness of social problem-solving therapy and reminiscence therapy as treatments for depression in older adults. J Consult Clin Psychol. 1993 Dec;61(6):1003-10. doi: 10.1037//0022-006x.61.6.1003. PMID 8113478
- [Background] Glasgow RE, Klesges LM, Dzewaltowski DA, Estabrooks PA, Vogt TM. Evaluating the impact of health promotion programs: using the RE-AIM framework to form summary measures for decision making involving complex issues. Health Educ Res. 2006 Oct;21(5):688-94. doi: 10.1093/her/cyl081. Epub 2006 Aug 31. PMID 16945984
- [Background] Glasgow RE, Strycker LA, King DK, Toobert DJ, Rahm AK, Jex M, Nutting PA. Robustness of a computer-assisted diabetes self-management intervention across patient characteristics, healthcare settings, and intervention staff. Am J Manag Care. 2006 Mar;12(3):137-45. PMID 16524346
- [Background] Fisher L, Mullan JT, Skaff MM, Glasgow RE, Arean P, Hessler D. Predicting diabetes distress in patients with Type 2 diabetes: a longitudinal study. Diabet Med. 2009 Jun;26(6):622-7. doi: 10.1111/j.1464-5491.2009.02730.x. PMID 19538238
- [Derived] Cashmore BA, Cooper TE, Evangelidis NM, Green SC, Lopez-Vargas P, Tunnicliffe DJ. Education programmes for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 Aug 22;8(8):CD007374. doi: 10.1002/14651858.CD007374.pub3. PMID 39171639
- [Derived] Hessler D, Fisher L, Glasgow RE, Strycker LA, Dickinson LM, Arean PA, Masharani U. Reductions in regimen distress are associated with improved management and glycemic control over time. Diabetes Care. 2014;37(3):617-24. doi: 10.2337/dc13-0762. Epub 2013 Oct 29. PMID 24170750
- [Derived] Fisher L, Hessler D, Glasgow RE, Arean PA, Masharani U, Naranjo D, Strycker LA. REDEEM: a pragmatic trial to reduce diabetes distress. Diabetes Care. 2013 Sep;36(9):2551-8. doi: 10.2337/dc12-2493. Epub 2013 Jun 4. PMID 23735726